CLINICAL TRIAL: NCT02882048
Title: A Randomized Controlled Trial of Auricular Acupuncture to Facilitate Outpatient Opioid Weaning
Brief Title: Auricular Acupuncture to Facilitate Outpatient Opioid Weaning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Heather Jackson, Assistant in Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160725
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Narcotic Addiction
Keywords: Opioid addiction; Opioid weaning
MeSH Terms: conditions — Narcotic-Related Disorders; Opioid-Related Disorders | interventions — Medication Therapy Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication management & NADA Protocol (Experimental): Standard of care medication management defined by opioid weaning protocol with specific, symptomatic medication regimens, and NADA protocol administered biweekly
  Interventions: Procedure: NADA Protocol; Other: Medication management
- Medication management (Active Comparator): Standard of care medication management defined by opioid weaning protocol with specific, symptomatic medication regimens.
  Interventions: Other: Medication management

INTERVENTIONS:
Procedure: NADA Protocol — NADA Protocol is a standardized acupuncture technique in which five designated points in the ear are needled.
  Other Names: National Acupuncture Detoxification Association Protocol
  Arms: Medication management & NADA Protocol
Other: Medication management — Standard of care medication management defined by an opioid weaning protocol with specific, symptomatic medication regimens.

SUMMARY:
This study is to compare two groups undergoing opioid weaning as ordered by their referring physicians. One group will undergo the standard opioid weaning process and the other group will have the addition of the NADA Protocol to the weaning process.

DETAILED DESCRIPTION:
The NADA (National Acupuncture Detoxification Association) Protocol is a standardized acupuncture technique in which five designated points in the ear are needled (+/-beads/seeds at points for home acupressure therapy in between treatments). The NADA Protocol is indicated for treatment of the following conditions: detoxification, withdrawal, emotional trauma, craving, stress syndromes, relapse prevention, rehabilitation & recovery maintenance. It is also commonly used for PTSD and addiction; however it has not been studied as an adjunct to outpatient opioid weaning protocols for pain.

It is cited in the literature as yielding improvements in engagement, retention, decreased cravings, anxiety, and physical symptoms. Given these documented results, it seems feasible the outpatient opioid weaning patient would likely benefit from this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Referral to the VUMC Interventional Pain Clinic for opioid weaning and discontinuation.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in clinical institute narcotic assessment scale (CINA) for withdrawal | time from beginning of opioid withdrawal intervention to opioid cessation(approximately 6 months)

SECONDARY OUTCOMES:
Off-opioids rate | time from beginning of opioid withdrawal intervention to opioid cessation(approximately 6 months)
Change from baseline assessment of psychological distress of weaning, assessed using the Hospital Anxiety and Depression Scale (HADS) | 9 months
Time to cessation of opioids | time from of beginning of opioid withdrawal intervention to opioid cessation (approximately 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jackson, MSN, APRN-BC, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson HJ, Walters J, Raman R. Auricular Acupuncture to Facilitate Outpatient Opioid Weaning: A Randomized Pilot Study. Med Acupunct. 2021 Apr 1;33(2):153-158. doi: 10.1089/acu.2020.1450. Epub 2021 Apr 19. PMID 33912273